CLINICAL TRIAL: NCT06817772
Title: Digital BIOmarkers for the Assessment of Motor Status in Parkinson's Disease Patients with CLInical and ThErapeutic Application
Acronym: BIOCLITE
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Asociación Parkinson Madrid (Other)
Responsible Party: Principal Investigator, Ignacio Pavón García, Associate Professor, Universidad Politecnica de Madrid
Other Study IDs: BDPLEDEMDP-IPG-DATOS-20231030; PID2021-123708OB-I00 (Other Grant/Funding Number: Spanish Ministry of Science and Innovation. Spanish State Research Agency)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Parkinson
Keywords: Parkinson; Biomarkers; Home monitoring; Wearable; Smartwatch
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's disease group: The inclusion criterion to this group is a diagnosis of Parkinson's disease based on the UK Brain Bank criteria.
- Healthy control group: The inclusion criterion is participants without movement disorders.

SUMMARY:
The goal of this observational study is to define digital biomarkers of motor symptoms in Parkinson's disease patients using wearable devices. The main questions it aims to answer is:

* Is there a biomarkers that allows the identification of PD from healthy controls?
* Is there a biomarkers that can identify the severity of the disease?
* Is there a biomarkers with clinical and therapeutic application that can be used in clinical and free living conditions to monitor the evolution of the disease?

Participants have to perform a set of guided exercises related to the MDS-UPDRS guide and daily living tasks, in supervised and unsupervised conditions.

DETAILED DESCRIPTION:
The participants must perform a set of exercises related to the MDS-UPDRS III scale and some free-living activities. These tasks must be performed wearing a smartwatch.

The activities will be done in supervised clinical and unsupervised free-living environments. The participants must perfom a baseline and a final assesment in supervised conditions and a week of free living monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease based on the UK Brain Bank criteria.
* Affiliated with Asociación Parkinson Madrid.
* Minimal or mild disease severity, defined by a Hoehn and Yahr scale score of ≤ 2.5.
* Be capable of performing the prescribed exercises independently.
* Maintain daily functioning without dependence on caregivers.

Exclusion Criteria:

* Hoehn and Yahr scale score of > 2.5.
* Have undergone deep brain stimulation, used dopamine infusion pumps, or have conditions mimicking PD symptoms (e.g., progressive supranuclear palsy, Lewy body dementia, multiple system atrophy, or other parkinsonian syndromes)
* Experience motor symptom fluctuations throughout the day.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the PD group, an initial and final evaluation will take place at the Asociación Parkinson Madrid. For the control group, the meeting will be at the Escuela Técnica Superior de Ingenieros Industriales at Universidad Politécnica de Madrid (ETSII-UPM).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for the identification of PD patients | 1 year
  A set of biomarkers will be defined for the identification of PD patients by comparing their data with that of healthy subjects.
biomarkers for the prediction MDS-UPDRS scores in PD patients | 1 year
  A collection of biomarkers will be calculated to predict MDS-UPDRS scores in PD patients
Biomarkers in supervised and unsupervised conditions | 1 year
  A comparation between the biomarkers defined in supervised settings versus those defined in free-living environments.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polvorinos-Fernández, C. et al. Evaluating Motor Symptoms in Parkinson's Disease Through Wearable Sensors: A Systematic Review of Digital Biomarkers. Appl. Sci. 2024, 14, 10189. https://doi.org/10.3390/app142210189
- [Background] Sigcha L, Polvorinos-Fernandez C, Costa N, Costa S, Arezes P, Gago M, Lee C, Lopez JM, de Arcas G, Pavon I. Monipar: movement data collection tool to monitor motor symptoms in Parkinson's disease using smartwatches and smartphones. Front Neurol. 2023 Dec 7;14:1326640. doi: 10.3389/fneur.2023.1326640. eCollection 2023. PMID 38148984
- [Derived] Polvorinos-Fernandez C, Sigcha L, Centeno-Cerrato M, de Arcas G, Grande M, Marin M, Parees I, Martinez-Castrillo JC, Pavon I. Evaluation of Free-Living Motor Symptoms in Patients With Parkinson Disease Through Smartwatches: Protocol for Defining Digital Biomarkers. JMIR Res Protoc. 2025 Jul 28;14:e72820. doi: 10.2196/72820. PMID 40720803
- See also: Related Info — http://i2a2.upm.es/bioclite